CLINICAL TRIAL: NCT03608956
Title: RENAL BLOOD FLOW MEASUREMENT WITH TRANSESOPHAGEAL ECHOCARDIOGRAPHY:RENAL OXYGEN SATURATION AND ITS ASSOCIATION WITH ACUTE RENAL INJURY
Brief Title: Renal Oxygen Saturation and Its Association With Acute Renal Injury
Status: Withdrawn | Type: Observational
Why Stopped: Withdrawn prior to recruitment due to institutional changes
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Mustafa Kemal Arslantas, Assoc. Prof. Dr, Marmara University
Other Study IDs: 09.2017.642
Record Dates: First submitted 2018-06-28; First posted 2018-08-01 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Acute Kidney Injury; Children; Cardiac Surgery
Keywords: regional oximetry; cerebral oximetry
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

SUMMARY:
Peri-operative renal dysfunction is a major mortality and morbidity cause following cardiac and major vascular surgery. Although several intra-operative strategies are proposed for better outcomes, no effective and fast resulting test is available to be done in operating rooms to assess renal functions. Urine and blood markers as serum creatinine, urine output, fractional excretion of sodium and urea are used for early diagnosis of acute renal injury. Near infrared spectroscopy (NIRS) assesses tissue oxygenation especially cerebral regional oxygen saturation. The benefit of NIRS followups of cerebral and somatic (liver, kidney, mesentery) oxygenation in pediatric cardiovascular surgery patients are demonstrated by studies.

DETAILED DESCRIPTION:
Peri-operative renal dysfunction is a major mortality and morbidity cause following cardiac and major vascular surgery. Patients undergoing cardiac surgery with more than one risk factor for postoperative renal insufficiency develop clinical significant renal dysfunction which results in extended length of stay in 1/5 of the patients .At least50% of the postoperative renal dysfunction is associated with development of renal hypoperfusion during cardiopulmonary bypass or aortic cross clamping. Although several intra-operative strategies are proposed for better outcomes, no effective and fast resulting test is available to be done in operating rooms to assess renal functions. Urine and blood markers as serum creatinine, urine output, fractional excretion of sodium and urea are used for early diagnosis of acute renal injury. In this study definition and classification of AKI (acute kidney injury) will be done according to KDIGO (kidney disease improving global outcome) criteria.

Renal perfusion can be assessed by renal artery measurements done by ultrasound imaging.The same assessment can also be done by transesophageal echocardiography (TEE).

Near infrared spectroscopy (NIRS) assesses tissue oxygenation especially cerebral regional oxygen saturation. NIRS measures regional oxygenation (rSO=oxyhemoglobin/ total Hemoglobin) by determining oxy- and deoxy- hemoglobin signals.

The probe placed on frontotemporal region has two sensors and a light source. Data is gained from sensors 3cm apart from the extracranial tissue and 4cm apart from the brain tissue; value is formed from calculation of the difference of these data. The benefit of NIRS followups of cerebral and somatic (liver, kidney, mesentery) oxygenation in pediatric cardiovascular surgery patients are demonstrated by studies.

The investigators aimed to investigate the association of postoperative acute renal injury and the change in peroperative renal blood flow and renal oxygenation values; additionally to establish wether it can be used as a fast responding and efficient method in evaluating renal function in the operating room settings.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients
* cardiovascular surgery
* Written informed consent
* Peroperative TEE assessment

Exclusion Criteria:

* Patients whose follow up cannot be done with TEE (ie Patients whose body weight is less than 5 kg, patients with esophageal pathologies)
* Patients with renal insufficiency

Patients whose TEE evaluation cannot be done optimally will be left out of the study

Ages: 1 Month to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients who meet the inclusion criteria and who will undergo cardiac surgery in our hospital will be included in the study.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-03-31 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
Early prediction of postoperative acute renal injury with TEE | Intraoperative period
  Intraoperative renal blood flow assessment with TEE
Early prediction of postoperative acute renal injury with transcutaneous renal regional oxygen saturation measured with NIRS | Intraoperative period
  Renal oxygenation values gained from NIRS monitor during the surgery
Acute kidney injury | Postoperative 1 week
  AKI is staged according to KDIGO

CONTACTS AND LOCATIONS:
Overall Officials: Alper Kararmaz, Prof, Principal Investigator — Marmara University Pendik Education and Research Hospital
Locations (1):
- Marmara University Pendik Education and Research Hospital, Istanbul, Turkey, Turkey (Türkiye)